CLINICAL TRIAL: NCT02993874
Title: Effect of Creatine Supplementation Associated to Clinical Treatment of the Functional Capacity of Patients With Intermittent Claudication.
Brief Title: Creatine Supplementation in Patients With Intermittent Claudication.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of Maringá (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Amazonas (Unknown)
Responsible Party: Principal Investigator, Ademar Avelar de Almeida Junior, PhD, State University of Maringá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Creatine PAD
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Intermittent Claudication
Keywords: Ergonemic resources; Walking capacity; Peripheral artery disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine (Experimental): Creatine monohydrate (Cr) Loading - 4 doses of 5g / day for 7 days Maintenance - 1 dose of 3g / day for 49 days Clinical treatment (30-45 minutes of walking, 3 times per week)
  Interventions: Dietary Supplement: Creatine
- Placebo (Placebo Comparator): Dextrose Loading - 4 doses of 5g / day for 7 days Maintenance - 1 dose of 3g / day for 49 days Clinical treatment (30-45 minutes of walking, 3 times per week)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine — The experimental group will ingest for seven days (Loading - phase 1), 5g (4x/day) of creatine monohydrate associated with the clinical treatment (30-45 minutes of walking, 3 times a week). Subsequently, they will ingest for 49 days (Maintenance - phase 2), 3g (1x / day) creatine monohydrate associated with clinical treatment (30-45 minutes of walking, 3 times a week). They will be given guidance by telephone, so that they can reach the necessary recommendations for the study.
  Other Names: Creatine and clinical treatment
  Arms: Creatine
Dietary Supplement: Placebo — The placebo group will ingest for seven days (Loading - phase 1), 5g (4x / day) of dextrose associated to clinical treatment (30-45 minutes of walking, 3 times per week). Subsequently, they will ingest for 49 days (Maintenance phase 2), 3g (1x / day) of dextrose associated with the clinical treatment (30-45 minutes of walking, 3 times a week). They will be given guidance by telephone, so that they can reach the necessary recommendations for the study.
  Other Names: Placebo and clinical treatment
  Arms: Placebo

SUMMARY:
The aim of this study will be to verify the effect of creatine supplementation associated to clinical treatment of the functional capacity in patients with intermittent claudication.

DETAILED DESCRIPTION:
The aim of this study will be to verify the effect of creatine supplementation associated to clinical treatment of the functional capacity in patients with intermittent claudication. The sample will be composed by patients with intermittent claudication of both sexes. The patients will be ramdomized in a double-blind procedure to receive during seven days (loading) and posteriorly 49 days (maintenance) a creatine (Cr) supplementation or placebo (PLA), associated to the clinical treatment. Before ("baseline"), after "loading" period and after the maintenance period of supplementation, the patients will go through a functional capacity evaluation. The fuctional capacity evaluation will be evaluated by a six minute-walking test. For statistical analysis it will be used the ANOVA of two factors for repeated measurements, having the (Cr and PLA) group and the time (pre, post-loading and post-maintenance), and when needed the post-hoc of Newman keuls. The adopted level of significance will be P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* symptom of pain during the six-minute walk test limited by leg pain due to intermittent claudication.
* present peripheral artery disease (Ankle-arm index < 0.90) in one or both limbs.
* Asymptomatic intermittent claudication determined from the clinical history.
* Not have muscle or joint injuries that make it impossible to practice physical activity.

Exclusion Criteria:

* not attending more than 15% of the intervention sessions or visits to the laboratory.
* Stick to a physical activity program in addition to that offered by the study.
* do not use medication regularly.
* aggravation of the disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change walking capacity | Baseline, one and eight weeks
  The walking capacity will be assessed through a six-minute walk test, before and after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA).

SECONDARY OUTCOMES:
Change oxygen saturation | Baseline, one and eight weeks
  Oxygen saturation will be assessed on calf region during the six-minute walk test through Near-infrared spectroscopy (NIRS, PortaMon, Artinis Medical Systems) before, after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA).
Change Short Physical Performance Battery | Baseline, one and eight weeks
  Functional capacity will be assessed through a Short Physical Performance Battery test, after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA).
Change cognitive function | Baseline, one and eight weeks
  For cognitive aspetcs evaluation the following procedures will be taken: Stroop test (Victoria Stroop test and N-Back (Operational Memory) will performed after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA).

OTHER OUTCOMES:
Change brachial blood pressure. | Baseline, one and eight weeks
  Brachial blood pressure will be assessed through an automatic monitor (HEM-742, Omron Healthcare, Japan) before, after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA).
Change arterial stiffness | Baseline, one and eight weeks
  The arterial stiffness will be evaluated by the applanation tonometry method (SphygmoCor, AtCor Medical, Australia) before, after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA).
Change autonomic cardiac modulation | Baseline, one and eight weeks
  The autonomic cardiac modulation will be evaluated through a heart rate monitor (Polar, RS 800, USA) after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA).
Change vasodilatory capacity | Baseline and eight weeks
  Vasodilatation capacity will be assessed by ultrasound imaging (HDI 5000 Sono CT, Philips, The Netherlands) after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups ( Cr and PLA).
Change body composition | Baseline and eight weeks
  Body composition will be evaluated after one week (Loading - 7 days) and after 7 weeks of supplementation (Maintenance - 49 days) in both groups (Cr and PLA) using the bio-electrical bioimpedance method (BIS 4200B Xitron Technologies, Inc, San Diego, PLA).
Creatine plasma | Baseline, one and eight weeks
  Creatine plasma will be evaluated by the High Performance Liquid Chromatography (HPLC) method (FL SPD-20A Shimadzu®, Kyoto, Japan), after one week (loading - 7 days) and after 7 weeks of supplementation (maintenance - 49 days) in both The groups (Cr and PLA).
Change of Renal function markers | Baseline, one and eight weeks
  serum creatinine,creatinine excretion rate and creatinine clearance. Urine will be collected during the 24-hour period, neglecting the first collection. For the measurement of the urinary volume, beakers of 500 to 1000 ml were used. Blood and urinary creatinine levels were determined by the Jaffé method without deproteinization.
Food habits | Baseline, one and eight weeks
  For food intake evaluation a 24-hour food diary will be required by previously trained nutritionists, using the nutritional evaluation program Avanutry 3.1.4

CONTACTS AND LOCATIONS:
Overall Officials: Ademar Avelar, PhD, Principal Investigator — State University of Maringa; Raphael Ritti-Dias, PhD, Study Director — Israel Institute of Education and Research Albert Einstein; Gabriel Cucato, PhD, Study Director — Israel Institute of Education and Research Albert Einstein
Locations (1):
- Israel Institute of Education and Research Albert Einstein, São Paulo, Brazil